CLINICAL TRIAL: NCT01665170
Title: A Randomized, Double Blind, Placebo-controlled Pilot Study on the Efficacy of Passiflora Incarnata L. in an Acute Stressful Situation
Brief Title: Pilot Study on the Efficacy of Pascoflair in an Acute Stressful Situation (TSST)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Collaborators: Daacro (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 178 S11 PF; 2011-006129-17 (EudraCT Number)
Record Dates: First submitted 2012-08-01; First posted 2012-08-15 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Healthy; Stress
Keywords: Pascoflair; tsst; passiflora incarnata; non smoking male; and female volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo
- Verum (Active Comparator): Verum arm - Pascoflair 425mg
  Interventions: Drug: Passiflora incarnata

INTERVENTIONS:
Drug: Passiflora incarnata — 3 x 1 tablet per day for 3 days
  Other Names: Pascoflair 425mg coated tablets
  Arms: Verum
Drug: Placebo — 3 x 1 ablet per day for 3 days
  Arms: Placebo

SUMMARY:
A randomized, double blind, placebo-controlled pilot study on the efficacy of Passiflora incarnata L. in an acute stressful situation

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, single-center study During Visit 1 study information and an informed consent form are handed out. After study inclusion on Visit 2, participants are assigned to one of two groups at random and receive the test products (either Pascoflair® or placebo tablets). The 3rd visit includes the completion of questionnaires regarding wellbeing and the Trier Social Stress Test.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent;
* Healthy male and female subjects
* Non-smoker;
* Age 25 to 45 years;
* BMI ≥ 19 to ≤ 30 kg/m2

Exclusion Criteria:

* Any known allergies to the test substance;
* Any known addiction to drugs, alcohol or positive results in the drug screening test;
* Any serious general illness, ongoing or within the last 12 months;
* Any febrile illness (> 24 hrs.) within 7 days prior to treatment;
* Any antibiotics for the last four weeks before study inclusion;
* Diabetes mellitus;
* Known heart disease, hypertension, kidney disease, significant respiratory disease, epilepsy, or rheumatoid arthritis;
* Known immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS) which could place the subject at risk or interfere with the accuracy of the study results;
* Pregnancy or lactating;
* Current participation or participation in any type of clinical study in the past week;
* Current or past participation in a TSST study;
* Employees of the Sponsor or the CRO;
* Any other medication that, in the opinion of the Investigator is likely to affect their response to treatment;
* Clinically relevant abnormalities in physical examinations, vital signs, clinical chemistry, or haematology as judged by the Investigator;
* Any other condition the Investigator or their duly assigned representatives believes may affect the ability of the individual to complete the study or the interpretation of the study results.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Clemens, MD, Prof, Principal Investigator — Klinikum Mutterhaus der Borromäerinnen GmbH, Feldstr. 16, 54290 Trier
Locations (1):
- Juliane Hellhammer, Trier, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals will be recruited via newspaper, mailing lists and radio advertisement in the area of Trier,Germany by DAaCRO. Recruiting: May 2012 - July 2012 in medical center/ CRO for Trier Social Sress Tests.
Pre-assignment Details: Three subjects were not included because the recruitment phase was already completed.
Groups:
- Placebo: Placebo arm, 3 x 1 tablet per every day for 3 days
- Verum: Verum arm - Pascoflair 425mg, 3 x 1 tablet per every day for 3 days
Period: Overall Study
Arm/Group | Placebo | Verum
Started | 30 (First patient in) | 30
Bevore TSST | 30 | 30
During TSST | 30 | 30
After TSST | 30 | 30
Completed | 30 (Last TSST/ last patient out) | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Verum | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.57 (5.00) | 28.47 (5.81) | 28.5 (5.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  Germany | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: VAS Insecurity (During)
Description: The primary objective is to assess effects of P. incarnata on psychological stress measured by Visual Analogue Scales (VAS; Bond and Lader 1974) by comparing scores collected before, during and after stress exposure between the P. incarnata and a placebo group. In this study, psychological stress is defined as stress perception, anxiety and insecurity. These three variables are determined simultaneously in the study before, during and after the stress test. Minimum = 0 mm; Maximum = 100 mm, higher value = represent a worsend outcome.
Time Frame: during stress test = Visite 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 30
mm | 56.87 (30.92) | 60.93 (30.39)

2. Primary Outcome: VAS Anxiety (During)
Description: as for outcome 1
Time Frame: during stress test = Visite 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Verum | Placebo
Number analyzed (Participants) | 30 | 30
mm | 29.67 (30.39) | 34.17 (30.92)

3. Secondary Outcome: Serum Cortisol (Pre-post Comparison)
Description: 2 min. prior to and 1 min. after the TSST
Time Frame: 1 day
Reporting Status: Not Posted

4. Secondary Outcome: ACTH (Pre-post Comparison)
Description: ACTH - Adrenocorticotropes Hormon - 2 min. prior to and 1 min. after the TSST
Time Frame: 1 day
Reporting Status: Not Posted

5. Secondary Outcome: Epinephrine (Before)
Description: 2 min. prior the TSST
Time Frame: 1 day
Reporting Status: Not Posted

6. Secondary Outcome: Norepinephrine (Before)
Description: 2 min. prior the TSST
Time Frame: before stress test
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 28 | 30
ng/dl | 430.29 (121.41) | 581.17 (160.82)

7. Secondary Outcome: State Anxiety (STAI-X1) Questionnaire
Description: The STAI-X1 measures state anxiety (one scale). Answers are given on a four-point rating scale ranging from 1 = "not at all" to 4 = "very true". The questionnaire is used as baseline measurement at V2. In addition, it is also employed before and immediately after the stress test at V3 to assess changes in state anxiety. Assess V2, before and after V3
Time Frame: 1 day
Reporting Status: Not Posted

8. Secondary Outcome: POMS Questionnaire
Description: The POMS assesses the four states depression/anxiety, fatigue, vigor and hostility (4 scales). High vigor scores reflect a positive mood whereas high scores in the other subscales indicate negative mood. Subjects rate their mood state on a 7-point rating scale ranging from 1 = "not at all" to 7 = "very strongly". The questionnaire is completed on V2 and V3.
Time Frame: 1 day
Reporting Status: Not Posted

9. Secondary Outcome: MDBF Questionnaire
Description: The MDBF assesses the three bipolar dimensions good/bad mood, wakefulness/tiredness and calmness/agitation (3 scales). The short form of the MDBF and its parallel version (versions A and B) each consist of 12 items. Subjects rate their mood state on a 5-point rating scale ranging from 1 = "not at all" to 5 = "very true". To determine mood changes induced by the TSST, the questionnaire is completed shortly before (version A) and immediately after the TSST (version B). Assess before and after V3
Time Frame: 1 day
Reporting Status: Not Posted

10. Secondary Outcome: LSEQ Questionnaire (Getting to Sleep-Falling Asleep Easier Than Usual) - Changes From V2 to V3
Description: The LSEQ investigates four aspects of sleep using VAS: getting to sleep, quality of sleep, awakening from sleep and behavior following awakening. The LSEQ is completed on V2 and V3.
  V2 = For each female, V2 is scheduled to take place on day 6 (-8) after the last contraceptive intake of a menstrual cycle. Upon arrival, subjects meeting all inclusion and no exclusion criteria are admitted to study participation and receive a random number starting from R001. V3 = After 2 days of treatment, the final appointment takes place in the afternoon. For each female, the appointment for V3 will be scheduled to take place on day 9 (-11) after the last contraceptive intake of a menstrual cycle. Females will be asked if oral contraceptives were administered on a regular basis and if pregnancy can be excluded. The LSEQ is a VAS scale 0 - 100mm, the value below is Change in percent; higher values represent a better outcome.
Time Frame: Visite 2 (before treatment), Visite 3 (after treatment)
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 29
Percent Change | 2.90 (24.23) | 11.21 (23.73)

11. Primary Outcome: VAS Stress Perception (During)
Description: as for outcome 1
Time Frame: during stress test = Visite 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 30
mm | 59.20 (28.77) | 57.3 (29.42)

12. Secondary Outcome: LSEQ Questionnaire (Getting to Sleep-Falling Asleep More Quickly Than Usual] - Changes From V2 to V3
Description: as for outcome 10
Time Frame: Visite 2 (before treatment), Visite 3 (after treatment)
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 30
Percent Change | 0.63 (25.78) | 11.47 (26.83)

13. Secondary Outcome: LSEQ Questionnaire (Getting to Sleep-Feeling More Drowsy Than Usual] - Changes From V2 to V3
Description: The LSEQ investigates four aspects of sleep using VAS: getting to sleep, quality of sleep, awakening from sleep and behavior following awakening. The LSEQ is completed on V2 and V3. V2 = For each female, V2 is scheduled to take place on day 6 (-8) after the last contraceptive intake of a menstrual cycle. Upon arrival, subjects meeting all inclusion and no exclusion criteria are admitted to study participation and receive a random number starting from R001. V3 = After 2 days of treatment, the final appointment takes place in the afternoon. For each female, the appointment for V3 will be scheduled to take place on day 9 (-11) after the last contraceptive intake of a menstrual cycle. Females will be asked if oral contraceptives were administered on a regular basis and if pregnancy can be excluded.
  The LSEQ is a VAS scale 0 - 100mm, the value below is Change in percent; lower values represent a better outcome.
Time Frame: Visite 2 (before treatment), Visite 3 (after treatment)
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 30
Percent Change | 3.67 (24.75) | -12.53 (23.35)

14. Secondary Outcome: LSEQ Questionnaire (Quality of Sleep - More Restful Than Usual] - Changes From V2 to V3
Description: as for outcome 10
Time Frame: Visite 2 (before treatment), Visite 3 (after treatment)
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 29
Percent Change | 1.53 (24.52) | 13.38 (26.81)

15. Secondary Outcome: LSEQ Questionnaire (Quality of Sleep - Fewer Periods of Wakefulness Than Usual] Changes From V2 to V3
Description: as for outcome 10
Time Frame: Visite 2, visite 3
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 29
Percent Change | 5.47 (27.80) | 14.59 (28.21)

16. Secondary Outcome: LSEQ Questionnaire (Awakening From Sleep- Easier Than Usual] Changes From V2 to V3
Description: as for outcome 10
Time Frame: Visite 2 (before treatment), Visite 3 (after treatment)
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 29
Percent Change | -0.33 (28.30) | 10.28 (27.23)

17. Secondary Outcome: LSEQ Questionnaire (Awakening From Sleep- Quicker Than Usual] Changes From V2 to V3
Description: as for outcome 10
Time Frame: Visite 2 (before treatment), Visite 3 (after treatment)
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 29
Percent Change | -6.07 (28.28) | 1.00 (29.64)

18. Secondary Outcome: LSEQ Questionnaire (Behavior Following Awakening- Feeling Alert Upon Awakening] Changes From V2 to V3
Description: as for outcome 10
Time Frame: Visite 2 (before treatment), Visite 3 (after treatment)
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 30
Percent Change | 5.63 (26.58) | 17.17 (23.90)

19. Secondary Outcome: LSEQ Questionnaire (Behavior Following Awakening- Feeling Alert Now] Changes From V2 to V3
Description: as for outcome 10
Time Frame: Visite 2 (before treatment), Visite 3 (after treatment)
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 29
Percent Change | 6.60 (32.92) | 19.17 (28.04)

20. Secondary Outcome: LSEQ Questionnaire (Behavior Following Awakening- Less Clumsy Balance and Coordination Upon Getting-up] Changes From V2 to V3
Description: The LSEQ investigates four aspects of sleep using VAS: getting to sleep, quality of sleep, awakening from sleep and behavior following awakening. The LSEQ is completed on V2 and V3. V2 = For each female, V2 is scheduled to take place on day 6 (-8) after the last contraceptive intake of a menstrual cycle. Upon arrival, subjects meeting all inclusion and no exclusion criteria are admitted to study participation and receive a random number starting from R001. V3 = After 2 days of treatment, the final appointment takes place in the afternoon. For each female, the appointment for V3 will be scheduled to take place on day 9 (-11) after the last contraceptive intake of a menstrual cycle. Females will be asked if oral contraceptives were administered on a regular basis and if pregnancy can be excluded.
  The LSEQ is a VAS scale 0 - 100mm, the value below is Change in percent; a higher value is a better outcome.
Time Frame: Visite 2 (before treatment), Visite 3 (after treatment)
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 29 | 30
Percent Change | -3.40 (16.53) | 1.66 (13.43)

21. Secondary Outcome: Norepinephrine (After)
Description: 2 min. after the TSST, higher value is better
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: ng/dl
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 28 | 29
ng/dl | 670.11 (204.61) | 803.14 (202.05)

22. Secondary Outcome: Sympathovagal Balance (Before TSST, Sitting - 1. Measurement)
Description: Sympathovagal balance is a measure of heart rate variability and gives information about the autonomic state that is regulated by sympathetic and parasympathetic influences. The low frequency component reflects sympathic activity, whereas the high requency domain gives Information about the parasympatic activity. Higher scores indicate a higher activation of the sympathic nervous System.
Time Frame: before TSST
Measure: Mean (Standard Deviation); unit: (low frequency/high frequency)*10
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 30
(low frequency/high frequency)*10 | 18.22 (7.66) | 22.84 (9.83)

23. Secondary Outcome: Sympathovagal Balance (Before TSST, Standing - 2. Measurement)
Description: as for outcome 22
Time Frame: before TSST
Measure: Mean (Standard Deviation); unit: (low frequency/high frequency)*10
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 29
(low frequency/high frequency)*10 | 27.74 (11.05) | 33.14 (13.89)

24. Secondary Outcome: Sympathovagal Balance (During TSST, Preparation - 3. Measurement)
Description: as for outcome 22
Time Frame: during TSST
Measure: Mean (Standard Deviation); unit: (low frequency/high frequency)*10
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 29
(low frequency/high frequency)*10 | 33.23 (12.21) | 38.37 (16.17)

25. Secondary Outcome: Sympathovagal Balance (During TSST, Interview - 4. Measurement)
Description: as for outcome 22
Time Frame: during TSST
Measure: Mean (Standard Deviation); unit: (low frequency/high frequency)*10
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 30
(low frequency/high frequency)*10 | 35.94 (13.94) | 39.25 (16.56)

26. Secondary Outcome: Sympathovagal Balance (During TSST, Arithmetics - 5. Measurement)
Description: as for outcome 22
Time Frame: during TSST
Measure: Mean (Standard Deviation); unit: (low frequency/high frequency)*10
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 30
(low frequency/high frequency)*10 | 44.01 (24.35) | 45.53 (20.23)

27. Secondary Outcome: Sympathovagal Balance (After TSST, Standing - 6. Measurement)
Description: as for outcome 22
Time Frame: after TSST
Measure: Mean (Standard Deviation); unit: (low frequency/high frequency)*10
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 30
(low frequency/high frequency)*10 | 42.36 (21.23) | 43.28 (17.71)

28. Secondary Outcome: Sympathovagal Balance (After TSST, Sitting - 7. Measurement)
Description: as for outcome 22
Time Frame: after TSST
Measure: Mean (Standard Deviation); unit: (low frequency/high frequency)*10
Arm/Group | Placebo | Verum
Number analyzed (Participants) | 30 | 30
(low frequency/high frequency)*10 | 26.42 (12.08) | 29.93 (13.35)

ADVERSE EVENTS:
Time Frame: 3 days (during the intake of the medication)
Arm/Group | Placebo | Verum
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No